CLINICAL TRIAL: NCT06682715
Title: Impact of Nutrition Education and Whey Supplementation on Body Composition and Endurance Performance of Athletes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Whey Supplementation
Record Dates: First submitted 2024-11-01; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: athlete; body composition; whey supplementation; endurance performance
MeSH Terms: interventions — Whey Proteins; maltodextrin; Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: A randomized study design will be used to compare the effects of whey vs maltodextrin (placebo) on university football players. The study will be performed during the time period of 7 weeks.In the 1st and 7th week, each participant will have their body composition analysed using InBody-270, USA. Parameters of interest in BIA are fat-mass, fat-free mass, BMI. Nutrition knowledge will be assessed using modified The Nutrition for Sports Knowledge Questionnaire and endurance performance will be assessed using Rockport fitness test (1mile test) / harvard step test for maximal oxygen calculation.
  Supplemental drinks will include 24g whey protein or iso-caloric amount of maltodextrin for placebo. Participants will be directed to perform their regular training sessions 5-6times/ week.
  Groups Dose Duration Treatment group(n=15) 24g whey protein 5 weeks Placebo group(n=15) Isocaloric maltodextrin 5 weeks
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whey group (Experimental): They will be given 24g of whey protein 5 days per week post workout.
  Interventions: Dietary Supplement: whey protein; Behavioral: nutrition education
- maltodextrin (Placebo Comparator): 35g of maltodextrin will be given 5 days per week post workout.
  Interventions: Dietary Supplement: maltodextrin; Behavioral: nutrition education

INTERVENTIONS:
Dietary Supplement: whey protein — 10 out of 20 participants will be randomly added in this group after initial consent in which they will be fully informed about all benefits, risks, and discomforts of this investigation. Screening process will include (1) subjects of age 18-30 years of age; (2) subjects should be free of any recent history of illnesses, musculoskeletal problems, and metabolic diseases; (3) are not using any supplements and medications; and (5) participated in ≥5 training sessions/week.
  Arms: whey group
Dietary Supplement: maltodextrin — 10 out of 20 participants will be randomly added in this group after initial consent in which they will be fully informed about all benefits, risks, and discomforts of this investigation. Screening process will include (1) subjects of age 18-30 years of age; (2) subjects should be free of any recent history of illnesses, musculoskeletal problems, and metabolic diseases; (3) are not using any supplements and medications; and (5) participated in ≥5 training sessions/week.
  Arms: maltodextrin
Behavioral: nutrition education — Nutrition for sports knowledge questionnaire will be used to assess the pre-nutrition education and post-nutrition education knowledge of athletes. Nutrition education will be given using evidence based nutrition education hand-outs and one-on-one counselling for each athlete in which they will be guided about sources of high biological value protein sources to meet daily protein requirement. Dietary intake will be monitored using 3 day food record method during 2-6 weeks of supplementation. Food logs will be filled out by participants during each weeks to monitor their protein intake. Three food logs (2 weekdays [Mon-Thurs/Tue-Fri] and 1 weekend day [Sat/Sun]) will be submitted by each subject every week.

SUMMARY:
Objectives of study are:

* Examining the influence of nutrition education/counseling on overall dietary protein consumption.
* Change in body composition parameters (body mass in kg, BMI kg/m2, fat mass(kg), fat free mass(kg), skeletal muscle mass(kg), percent body fat ) measured by InBody-270 analyzer over 5 weeks.
* Change in maximal oxygen consumption assessed using the Rockport Fitness Test after 5 weeks of supplementation.

  20 participants will be randomly assigned to whey or placebo (maltodextrin) group. Pre and post-analysis will be done for body composition, nutrition knowledge and dietary assessment and maximal oxygen consumption. Along with supplementation during week 2-6, individualized nutrition education with food logging will be provided with their programmed training. Changes in body composition (body mass in kg, BMI kg/m2, fat mass(kg), fat free mass(kg), skeletal muscle mass(kg), percent body fat) using In Body Composition Analyzer, maximal oxygen consumption using Rockport Fitness test (1 mile test), protein intake and nutrition knowledge using Nutrition for Sports Knowledge Questionnaire will be assessed.

DETAILED DESCRIPTION:
Proposed place of work:

I. Football team players from public universities in Lahore.

Plan of work and methodology adopted:

* Study design: Experimental
* Duration of study: 7 weeks
* Participants recruitment: 20 male football players, aged between 18-30 years.

Intervention plan:

Groups Dose Duration Treatment group(n=15) 24g whey protein 5 weeks Placebo group(n=15) Isocaloric maltodextrin 5 weeks

Subjects:

Participants (n=20) will be recruited after initial consent in which they will be fully informed about all benefits, risks, and discomforts of this investigation. Screening process will include Minimum Age: 18 Years Maximum Age: 30 Years

Inclusion Criteria:

Age range: 18-30 years BMI: 18.5 kg/m² to 30 kg/m² Participation in ≥5 training sessions per week

Exclusion Criteria:

Known allergies to whey Recent history of illnesses, musculoskeletal issues, or metabolic diseases use supplementation/medication

Research layout plan:

A randomized study design will be used to compare the effects of whey vs maltodextrin (placebo) on university football players. The study will be performed during the time period of 7 weeks.

Pre and post testing:

In the 1st and 7th week, each participant will have their body composition analysed using InBody-270, USA. Parameters of interest in BIA are fat-mass, fat-free mass, BMI. Nutrition knowledge will be assessed using modified The Nutrition for Sports Knowledge Questionnaire and endurance performance will be assessed using Rockport fitness test (1mile test) for maximal oxygen consumption calculation.

Dietary assessment:

3 day food dietary recall will be used initially in the 1st week to assess their dietary protein intake. Based on a dietary analysis, participants will be given a dietary plan (taking into account the resting metabolic rate and total daily physical activity related energy expenditure) and their daily protein needs will be calculated using 1.4g/kg of body weight for each participant.

Nutrition education and supplementation:

Nutrition education will be given using evidence based nutrition education hand-outs and one-on-one counselling for each athlete in which they will be guided about sources of high biological value protein sources to meet daily protein requirement. Dietary intake will be monitored using 3 day food record method during 2-6 weeks of supplementation. Food logs will be filled out by participants during each week to monitor their protein intake. Three food logs (2 weekdays [Mon-Thurs/Tue-Fri] and 1 weekend day [Sat/Sun]) will be submitted by each subject every week.

Supplemental drinks will include 24g whey protein or iso-caloric amount of maltodextrin for placebo. Participants will be directed to perform their regular training sessions 5-6times/ week.

Performance test:

A valid field test to determine maximal oxygen consumption in the public is the Rockport Walk Fitness test. Furthermore, it requires little preparation and can be delivered to big crowds. Participants will be given instructions to abstain from strenuous exercise beginning 24 hours before to Rockport walk/run fitness test. On the day of the exam, they will be instructed to eat a light breakfast and report to the gym for recording after two hours. On the treadmill, participants will be told to walk as quickly as they can for 1 mile. The stopwatch will be used to time how long it takes to finish the test. The heart rate will be assessed pre and post 1 mile walk. Maximal oxygen consumption will be calculated by using equation.

ELIGIBILITY:
Inclusion Criteria:

* Age (18-35)Individuals with BMI ranging from 18.5 kg/m2 to 30 kg/m2
* participated in ≥5 training sessions/week

Exclusion Criteria:

* Individuals who have any known allergies especially whey
* any recent history of illnesses, musculoskeletal problems, and metabolic diseases

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — biological male
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-03-22 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in body composition parameters (% fat mass, % fat-free mass, BMI) measured by InBody-270 analyzer over 5 weeks | 5 weeks
  after 5 weeks of supplementation parameters like %fat-mass, %fat-free mass and BMI improve.
Change in maximal oxygen consumption (VO2 max) assessed using the Rockport Fitness Test after 5 weeks of supplementation | 5 weeks
  after 5 weeks of supplementation, maximal oxygen consumption will increase

SECONDARY OUTCOMES:
Change in dietary protein intake measured by 24-hour dietary recall and 3-day food records over the 5-week intervention. | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: waqas ahmad, Study Chair — Associate Professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang WC, Chang YC, Chen YM, Hsu YJ, Huang CC, Kan NW, Chen SS. Whey Protein Improves Marathon-Induced Injury and Exercise Performance in Elite Track Runners. Int J Med Sci. 2017 Jun 22;14(7):648-654. doi: 10.7150/ijms.19584. eCollection 2017. PMID 28824296
- [Result] Taylor LW, Wilborn C, Roberts MD, White A, Dugan K. Eight weeks of pre- and postexercise whey protein supplementation increases lean body mass and improves performance in Division III collegiate female basketball players. Appl Physiol Nutr Metab. 2016 Mar;41(3):249-54. doi: 10.1139/apnm-2015-0463. Epub 2015 Nov 9. PMID 26842665
- [Result] Poulios A, Fatouros IG, Mohr M, Draganidis DK, Deli C, Papanikolaou K, Sovatzidis A, Nakopoulou T, Ermidis G, Tzatzakis T, Laschou VC, Georgakouli K, Koulouris A, Tsimeas P, Chatzinikolaou A, Karagounis LG, Batsilas D, Krustrup P, Jamurtas AZ. Post-Game High Protein Intake May Improve Recovery of Football-Specific Performance during a Congested Game Fixture: Results from the PRO-FOOTBALL Study. Nutrients. 2018 Apr 16;10(4):494. doi: 10.3390/nu10040494. PMID 29659539
- [Result] Jenner SL, Buckley GL, Belski R, Devlin BL, Forsyth AK. Dietary Intakes of Professional and Semi-Professional Team Sport Athletes Do Not Meet Sport Nutrition Recommendations-A Systematic Literature Review. Nutrients. 2019 May 23;11(5):1160. doi: 10.3390/nu11051160. PMID 31126159